CLINICAL TRIAL: NCT06118957
Title: A Pilot Randomized Controlled Trial of Low Molecular Weight Heparin or no Treatment Following Cesarean Delivery
Brief Title: Low Molecular Weight Heparin or no Treatment Following Cesarean Delivery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Ann Bruno, Assistant Professor Obstetrics And Gynecology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00167480
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Thromboembolism
Keywords: Thromboembolism; Enoxaparin; Cesarean delivery
MeSH Terms: conditions — Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enoxaparin (Experimental): Participants will receive weight-based dosing of enoxaparin at 0.5 mg/kg rounded to the nearest 10 mg every 12 hours based on delivery admission weight. Participants will receive therapy for 14 days.
  Interventions: Drug: Enoxaparin
- No treatment (No Intervention): Participants will receive no enoxaparin treatment.

INTERVENTIONS:
Drug: Enoxaparin — Participants will receive weight-based dosing of enoxaparin at 0.5 mg/kg rounded to the nearest 10 mg every 12 hours based on delivery admission weight. Participants will receive therapy for 14 days.
  Arms: Enoxaparin

SUMMARY:
The aim of this study is to evaluate the feasibility of randomizing individuals to low molecular weight heparin (enoxaparin) or no treatment following cesarean delivery. The investigators hypothesize that among eligible individuals, at least 35% will enroll, undergo randomization, and complete the allocated treatment group.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a major contributor to maternal morbidity and mortality. The first two weeks postpartum are the highest risk period for VTE during pregnancy and the postpartum period. Cesarean delivery is a known risk factor for VTE. In the United States, postpartum prophylaxis with low molecular weight heparin (e.g., enoxaparin) is commonly used during the first 10-14 days after delivery. Enoxaparin has not been demonstrated as an effective intervention to prevent postpartum VTE after cesarean delivery. Before larger scale studies may be completed, a better understanding of ability to randomize individuals to this intervention is needed. This study aims to evaluate the feasibility of randomizing individuals after cesarean delivery to the receipt of enoxaparin prophylaxis or no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery at the University of Utah Health

Exclusion Criteria:

* Contraindication to anticoagulation
* Plan for therapeutic anticoagulation
* Known renal dysfunction (creatinine clearance <30mL/minute)
* History of venous thromboembolism
* High risk thrombophilia
* Receipt of antepartum anticoagulation for >2 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Bruno, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Enoxaparin: Participants will receive weight-based dosing of enoxaparin at 0.5 mg/kg rounded to the nearest 10 mg every 12 hours based on delivery admission weight. Participants will receive therapy for 14 days
- No Intervention: No Treatment: Participants will receive no enoxaparin treatment.
Period: Overall Study
Arm/Group | Experimental: Enoxaparin | No Intervention: No Treatment
Started | 32 | 32
Completed | 32 | 29
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: Rate of approach and enrollment of all screened eligible patients over the six-month study period by month
Groups:
- Enrolled: Participants who enrolled in the study
- Declined: Patients who declined participation in the study
- Total: Total of all reporting groups
Arm/Group | Enrolled | Declined | Total
Number analyzed (Participants) | 64 | 547 | 611
Age, Continuous [Median (Standard Deviation); unit: years of age] | 30.95 (5.5) | 31.37 (5.7) | 31.32 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 547 | 611
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 156 | 170
  Not Hispanic or Latino | 40 | 315 | 355
  Unknown or Not Reported | 10 | 76 | 86

OUTCOME MEASURES:

1. Primary Outcome: Rate of Eligible Individuals Enrolled and Retained Through Full Study Procedures
Description: Feasibility as defined by ≥35% enrollment of eligible individuals and retention ≥85% of enrolled individuals through all study procedures
Time Frame: A pilot randomized controlled trial of low molecular weight heparin or no treatment following cesarean delivery NCT06118957 July 30, 2025 6 weeks
Measure: Number; unit: participants
Groups:
- Eligible Participants: Eligible Participants for Enrollment in the Study
Arm/Group | Eligible Participants
Number analyzed (Participants) | 694
participants
  # of eligible patients | 694
  Approach rate (proportion of eligible patients approached) | 611
  Enrollment rate (proportion of eligible patients enrolled) | 64
  Retention rate (proportion enrolled completing study) | 61

2. Secondary Outcome: Rate of Venous Thromboembolism
Description: Objectively (by imaging) diagnosed deep vein thrombosis or pulmonary embolism
Time Frame: 6 Weeks
Population: There were no reported incidents for venous thromboembolism
Measure: Number; unit: # of venous thromboembolism events
Arm/Group | Enoxaparin | No Treatment
Number analyzed (Participants) | 32 | 32
# of venous thromboembolism events | 0 | 0

3. Secondary Outcome: Rate of Wound Hematoma or Infection
Description: Clinically diagnosed
Time Frame: 6 Weeks
Measure: Number; unit: # of reported wound hematoma events
Arm/Group | Experimental: Enoxaparin | No Intervention: No Treatment
Number analyzed (Participants) | 32 | 32
# of reported wound hematoma events | 2 | 1

4. Secondary Outcome: Rate of Bleeding Complications
Description: Clinically diagnosed as readmission to hospital for bleeding or delayed postpartum hemorrhage (>24 hours after delivery)
Time Frame: 6 Weeks
Measure: Number; unit: # of reported bleeding complication even
Arm/Group | Experimental: Enoxaparin | No Intervention: No Treatment
Number analyzed (Participants) | 32 | 32
# of reported bleeding complication even | 0 | 1

ADVERSE EVENTS:
Time Frame: Within 6 Weeks Postpartum
Description: Complications by study group
Groups:
- No Treatment-: Participants will receive no enoxaparin treatment.
Arm/Group | Enoxaparin | No Treatment-
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 4/32 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoxaparin (N=32) | No Treatment- (N=32)
Blood in Breast Milk (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Patient concern for blood in breast milk. Clinician examination negative and concern resolved.
cholelithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Presentation to emergency department with right upper quadrant pain. Labs and ultrasound obtained consistent with cholelithiasis. Discharged with oral pain regimen.
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — Superficial surgical site infection with cellulitis, treated with oral antibiotics.
Uterine Rupture with broad ligament hematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — uterine rupture with broad ligament expanding hematoma requiring return to surgery on post day # for evacuation of hemoperitoneum. Patient enrolled in trial but not yet received therapy or no therapy per randomization (at clinician discretion).
Surgical site infection (Infections and infestations) | 1 (1) | 0 (0) — Surgical site infection with abscess requiring intravenous antibiotics and incision drainage.
Superficial incision separation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Superficial incision separation (2 mm by clinician examination).
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Presentation to emergency department with right upper quadrant pain. Labs and imaging obtained consistent with acute idiopathic pancreatitis without necrosis or infection. Conservatively managed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT06118957/Prot_SAP_ICF_002.pdf